CLINICAL TRIAL: NCT05993663
Title: Museums as Health Spaces: Design and Evaluation of the Effectiveness of an Arts in Health Intervention to Improve the Quality of Life and Functional Capacity Regarding the Pain of People With Fibromyalgia. Mixed Methodology Study.
Brief Title: Effectiveness of an Intervention Based on Arts In Health in the Quality of Life of People With Fibromyalgia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Agència de Salut Pública de Catalunya (ASPCAT) (Unknown); Institut Català de la Salut (Other); Servei de Museus i Protecció de Béns Mobles (Unknown); Museu de l'Empordà (Unknown); Adhoc Cultura (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23/133-P
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Arts in Health; Mindfulness; Visual Thinking Strategies; Revised Fibromyalgia Impact Questionnaire (FIQ-R)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Single intervention will be carried out for the 60 people who are part of the intervention groups, which will be 4 in total
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention groups that will receive 12 Arts in Health session. There will be four groups of 15 individuals for reaching the needed sample size.
  Interventions: Behavioral: Arts in health group intervention
- Control group (No Intervention): Control groups. Participants in these groups won't receive any group intervention, just regular health care.

INTERVENTIONS:
Behavioral: Arts in health group intervention — 12 sessions using the Arts in Health methodology with the aim of having a better understanding of the disease, developing healthy lifestyle habits and greater emotional intelligence. Visual thinking strategies, game based activities, mindfulness and dance will be used
  Arms: Intervention group

SUMMARY:
The aim of this intervention is to measure the impact of a 12-session intervention with Arts in Health methodology on the quality of life of the population with fibromyalgia.

The main questions it aims to answer are:

* To know if the methodology of Arts in Health is effective for the improvement of the functional capacity of people with fibromyalgia
* Which are the most effective techniques within this intervention

During the intervention, the participants will take part in mindfulness sessions, dance, visual thinking strategies, aimed at a greater understanding of the disease and the development of healthy habits.

The results of this intervention are compared with a control group, in which the same scales and instruments will be passed in the same period of time. To complete the information gathering, a focus group will be held to obtain qualitative information about the experience of the participants.

DETAILED DESCRIPTION:
Arts in Health is a methodology that seeks to use the power of arts and culture to improve people's health and well-being. To develop it, collaboration is promoted between health professionals and those in the artistic and cultural fields.

In accordance with the Arts in Health strategy of the Catalan Health Institute, the primary health care professionals in Figueres have started a joint project along Museu de l'Empordà, a local museum, to address fibromyalgia from this perspective.

The objectives are to quantitatively analyze the effectiveness of an Arts in Health intervention to improve the functional capacity with respect to pain and the quality of life of people with fibromyalgia. Also, qualitatively assess the experience of the participants and explore how they value the impact of cultural activities on health.

Joint work has been carried out to produce a guide where, through different modalities of Art, the symptoms and needs of people suffering from fibromyalgia will be addressed. Affected people have also collaborated in this process. With the results of this work, the content of the Intervention has been designed.

From here, a mixed methodology study is proposed through a randomized clinical trial for people affected by fibromyalgia. For the quantitative analysis, quality of life tests and a disability perception test due to pain, (FIQ-R), will be taken before, at the end and 6 months after the intervention. For the qualitative analysis, focus groups will be formed at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with fibromyalgia (M79.1) or diagnosed with fibromyalgia and chronic fatigue syndrome (T78.40 and M79.7)
2. Over 18 years old.
3. They agree to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Serious concomitant rheumatological pathology, that is to say, that this involves a much more important functional disability than that caused by the fibromyalgia pathology itself.
2. Serious psychiatric pathology [according to V Diagnostical and Statical Manual of Mental Disorders (DSM-V) criteria] that could make it difficult to participate in the sessions and follow the study. Or that due to his psychiatric diagnosis, participation in a group was not advisable because of the negative impact it could cause.
3. Having previously participated in the group education project for people with fibromyalgia in Figueres Health Care Center.
4. Users who present a language barrier that makes good communication impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | The first and last days of the intervention and 6 months after intervention.
  Functional capacity with respect to pain management, measured with the Revised Fibromyalgia Impact Questionnaire (FIQ-R)
Life quality | The first and last days of the intervention and 6 months after intervention.
  Quality of life perceived by the participants, measured with the EUROQOL

SECONDARY OUTCOMES:
Anxiety | 1 month before the intervention, last intervention day and 6 months after intervention.
  Assessment of anxiety with the Goldberg scale
Emotional well-being | 1 month before the intervention, last intervention day and 6 months after intervention.
  Assessment of emotional well-being with the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS)
Depression | 1 month before the intervention, last intervention day and 6 months after intervention.
  Depression
Social support | 1 month before the intervention, last intervention day and 6 months after intervention.
  Assessment of perceived social support with the Oslo Social Support Scale (OSLO-3) scale
Drug consumption | During the 6 months before the intervention and the 6 months after the intervention.
  Painkillers and psychotropic drugs consumed
Health care professional appointments. | During the 6 months before the intervention, during the interventions and the 6 months after the intervention.
  Assistance to health services

CONTACTS AND LOCATIONS:
Locations (1):
- ABS Figueres, Figueres, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bravo C, Skjaerven LH, Guitard Sein-Echaluce L, Catalan-Matamoros D. Effectiveness of movement and body awareness therapies in patients with fibromyalgia: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2019 Oct;55(5):646-657. doi: 10.23736/S1973-9087.19.05291-2. Epub 2019 May 15. PMID 31106558
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Bellato E, Marini E, Castoldi F, Barbasetti N, Mattei L, Bonasia DE, Blonna D. Fibromyalgia syndrome: etiology, pathogenesis, diagnosis, and treatment. Pain Res Treat. 2012;2012:426130. doi: 10.1155/2012/426130. Epub 2012 Nov 4. PMID 23213512
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Glombiewski JA, Sawyer AT, Gutermann J, Koenig K, Rief W, Hofmann SG. Psychological treatments for fibromyalgia: a meta-analysis. Pain. 2010 Nov;151(2):280-295. doi: 10.1016/j.pain.2010.06.011. Epub 2010 Aug 19. PMID 20727679
- [Background] Bernardy K, Fuber N, Kollner V, Hauser W. Efficacy of cognitive-behavioral therapies in fibromyalgia syndrome - a systematic review and metaanalysis of randomized controlled trials. J Rheumatol. 2010 Oct;37(10):1991-2005. doi: 10.3899/jrheum.100104. Epub 2010 Aug 3. PMID 20682676
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Mayorga Buiza, M. J. et al. Impacto de un programa de educación sanitaria en pacientes con fibromialgia. Rev. la Soc. Española del Dolor 17, 227-232 (2010).
- [Background] García-Campayo, J. et al. Intervención psicoeducativa en pacientes con fibromialgia en Atención Primaria: Efectividad y diferencias entre terapia individual y grupal. Cuad. Med. Psicosomática 73, 32-41 (2005)
- [Background] van Koulil S, Effting M, Kraaimaat FW, van Lankveld W, van Helmond T, Cats H, van Riel PL, de Jong AJ, Haverman JF, Evers AW. Cognitive-behavioural therapies and exercise programmes for patients with fibromyalgia: state of the art and future directions. Ann Rheum Dis. 2007 May;66(5):571-81. doi: 10.1136/ard.2006.054692. Epub 2006 Aug 17. PMID 16916856
- [Background] Drozd M, Marzęda M, Blicharz A, Czarnota J, Piecewicz-Szczęsna H. Unclear etiology and current hypotheses of the pathogenesis of fibromyalgia. J Educ Health Sport [Internet]. 2020 Sep. 15 [cited 2023 Jun. 8];10(9):338-44.
- [Background] Daykin, N. (2016). Arts for Health and Wellbeing. An Evaluation Framework.
- [Background] Fancourt D, Finn S. What is the evidence on the role of the arts in improving health and well-being? A scoping review [Internet]. Copenhagen: WHO Regional Office for Europe; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK553773/ PMID 32091683
- [Background] Clift S, Camic PM. Oxford Textbook of Creative Arts, Health, and Wellbeing: International Perspectives on Practice, Policy, and Research. Oxford: Oxford University Press; 2016
- [Background] Siles S, Castillejo M, Fernández J, Larraín A, Azcona C. Prácticas artísticas en contextos de salud comunitaria: cinco experiencias de arte y salud en los Centros Municipales de Salud Comunitaria de Madrid. Arteterapia [Internet]. 2020 [consultat el 07 de març de 2023]; 15: 135-146. Avaliable at: https://revistas.ucm.es/index.php/ARTE/article/view/65388/4564456554480
- [Background] Staricoff RL. Arts in Health: a review of the medical literature. Arts Council England; 2004. Available at: http://archive.artsandhealth.org/public/Resources/Research%20MedLitReview%20Dr%20Staricoff.pdf
- [Background] Montse Grifoll et al. Museus i Salut, Generalitat de Catalunya. Departament de Salut.2022
- [Background] Baptista AS, Villela AL, Jones A, Natour J. Effectiveness of dance in patients with fibromyalgia: a randomized, single-blind, controlled study. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):18-23. Epub 2012 Dec 14. PMID 23020850
- [Background] Hickman B, Pourkazemi F, Pebdani RN, Hiller CE, Fong Yan A. Dance for Chronic Pain Conditions: A Systematic Review. Pain Med. 2022 Dec 1;23(12):2022-2041. doi: 10.1093/pm/pnac092. PMID 35736401
- [Background] Murillo-Garcia A, Villafaina S, Adsuar JC, Gusi N, Collado-Mateo D. Effects of Dance on Pain in Patients with Fibromyalgia: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2018 Oct 1;2018:8709748. doi: 10.1155/2018/8709748. eCollection 2018. PMID 30364046
- [Background] Fancourt D. Arts in Health: Designing and Researching Interventions. Oxford University Press; 2017
- [Background] Warran K, Burton A, Fancourt D. What are the active ingredients of 'arts in health' activities? Development of the INgredients iN ArTs in hEalth (INNATE) Framework. Wellcome Open Res. 2022 Apr 29;7:10. doi: 10.12688/wellcomeopenres.17414.2. eCollection 2022. PMID 35600003
- [Background] Staricoff RL. Arts in Health: a review of the medical literature. Arts Council England; 2004
- [Background] Lloyd J, Barz G, Brummel-Smith K. The Oxford Handbook of Medical Ethnomusicology. Oxford University Press; 2008.
- [Background] Poulos RG, Marwood S, Harkin D, Opher S, Clift S, Cole AMD, Rhee J, Beilharz K, Poulos CJ. Arts on prescription for community-dwelling older people with a range of health and wellness needs. Health Soc Care Community. 2019 Mar;27(2):483-492. doi: 10.1111/hsc.12669. Epub 2018 Oct 21. PMID 30345578
- [Background] Salgueiro M, Garcia-Leiva JM, Ballesteros J, Hidalgo J, Molina R, Calandre EP. Validation of a Spanish version of the Revised Fibromyalgia Impact Questionnaire (FIQR). Health Qual Life Outcomes. 2013 Aug 1;11:132. doi: 10.1186/1477-7525-11-132. PMID 23915386
- [Background] Perez-Aranda A, Andres-Rodriguez L, Feliu-Soler A, Nunez C, Stephan-Otto C, Pastor-Mira MA, Lopez-Roig S, Penacoba C, Calandre EP, Slim M, Salgueiro M, Feixas G, Luciano JV. Clustering a large Spanish sample of patients with fibromyalgia using the Fibromyalgia Impact Questionnaire-Revised: differences in clinical outcomes, economic costs, inflammatory markers, and gray matter volumes. Pain. 2019 Apr;160(4):908-921. doi: 10.1097/j.pain.0000000000001468. PMID 30586023
- [Background] Luciano JV, Aguado J, Serrano-Blanco A, Calandre EP, Rodriguez-Lopez CM. Dimensionality, reliability, and validity of the revised fibromyalgia impact questionnaire in two Spanish samples. Arthritis Care Res (Hoboken). 2013 Oct;65(10):1682-9. doi: 10.1002/acr.22034. PMID 23609980
- [Background] Sandiumenge, L. Catalunya entoma la fibromiàlgia i la fatiga crònica. Act. Parlam. (2008)
- [Background] Guia per a l'avaluació de la fibromiàlgia i de la síndrome de fatiga crònica. Generalitat de Catalunya Departament de Salut
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Background] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Background] Monterde, S. Validación de la versión española del Fibromyalgia Impact Questionnaire. Rev. española Reumatol. Órgano Of. la Soc. Española Reumatol. 2004; 31, 507.
- [Background] Koebner IJ, Bonilla B, Slatman J, Parry M. The Analgesic Museum. Front Pain Res (Lausanne). 2022 Oct 21;3:1019632. doi: 10.3389/fpain.2022.1019632. eCollection 2022. PMID 36341154
- [Background] Koebner IJ, Chatterjee HJ, Tancredi DJ, Witt CM, Gosdin M, Rawal R, Weinberg G, Meyers FJ. Developing a framework for arts in health programs targeting individuals with chronic pain: a mixed-methods study of practitioners. Public Health. 2021 Aug;197:68-74. doi: 10.1016/j.puhe.2021.05.032. Epub 2021 Aug 3. PMID 34352682
- [Background] Barrenengoa-Cuadra MJ, Angon-Puras LA, Moscosio-Cuevas JI, Gonzalez-Lama J, Fernandez-Luco M, Gracia-Ballarin R. [Effectiveness of pain neuroscience education in patients with fibromyalgia: Structured group intervention in Primary Care]. Aten Primaria. 2021 Jan;53(1):19-26. doi: 10.1016/j.aprim.2019.10.007. Epub 2020 Feb 6. Spanish. PMID 32033824
- [Background] Thomson LJ, Lockyer B, Camic PM, Chatterjee HJ. Effects of a museum-based social prescription intervention on quantitative measures of psychological wellbeing in older adults. Perspect Public Health. 2018 Jan;138(1):28-38. doi: 10.1177/1757913917737563. Epub 2017 Nov 13. PMID 29130869
- [Background] Fontaine KR, Conn L, Clauw DJ. Effects of lifestyle physical activity on perceived symptoms and physical function in adults with fibromyalgia: results of a randomized trial. Arthritis Res Ther. 2010;12(2):R55. doi: 10.1186/ar2967. Epub 2010 Mar 30. PMID 20353551
- [Background] Martin L, Oepen R, Bauer K, Nottensteiner A, Mergheim K, Gruber H, Koch SC. Creative Arts Interventions for Stress Management and Prevention-A Systematic Review. Behav Sci (Basel). 2018 Feb 22;8(2):28. doi: 10.3390/bs8020028. PMID 29470435
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Macnaughton J, Stephen AI, Fleming MJ. The creative arts in palliative care. Oxford Research Encyclopedia of Communication; 2017
- [Background] Stuckey HL, Nobel J. The connection between art, healing, and public health: a review of current literature. Am J Public Health. 2010 Feb;100(2):254-63. doi: 10.2105/AJPH.2008.156497. Epub 2009 Dec 17. PMID 20019311
- [Background] Bosman JT, Bood ZM, Scherer-Rath M, Dorr H, Christophe N, Sprangers MAG, van Laarhoven HWM. The effects of art therapy on anxiety, depression, and quality of life in adults with cancer: a systematic literature review. Support Care Cancer. 2021 May;29(5):2289-2298. doi: 10.1007/s00520-020-05869-0. Epub 2020 Nov 13. PMID 33188476
- [Background] Young R, Camic PM, Tischler V. The impact of community-based arts and health interventions on cognition in people with dementia: a systematic literature review. Aging Ment Health. 2016;20(4):337-51. doi: 10.1080/13607863.2015.1011080. Epub 2015 Feb 16. PMID 25683767
- [Background] Onieva-Zafra MD, Castro-Sanchez AM, Mataran-Penarrocha GA, Moreno-Lorenzo C. Effect of music as nursing intervention for people diagnosed with fibromyalgia. Pain Manag Nurs. 2013 Jun;14(2):e39-46. doi: 10.1016/j.pmn.2010.09.004. Epub 2010 Nov 26. PMID 23108015
- [Background] Macnaughton, J., White, M., & Stacy, R. Researching the benefits of Arts in Health. Health Education, 2005; 105(5), 332-339.
- [Background] Camic PM, Baker EL, Tischler V. Theorizing How Art Gallery Interventions Impact People With Dementia and Their Caregivers. Gerontologist. 2016 Dec;56(6):1033-1041. doi: 10.1093/geront/gnv063. Epub 2015 Jul 16. PMID 26185152
- [Background] Daykin N, Mansfield L, Meads C, Julier G, Tomlinson A, Payne A, Grigsby Duffy L, Lane J, D'Innocenzo G, Burnett A, Kay T, Dolan P, Testoni S, Victor C. What works for wellbeing? A systematic review of wellbeing outcomes for music and singing in adults. Perspect Public Health. 2018 Jan;138(1):39-46. doi: 10.1177/1757913917740391. Epub 2017 Nov 13. PMID 29130840